CLINICAL TRIAL: NCT00602355
Title: Placebo Controlled Trial of Sertraline and Interpersonal Psycho-Therapy for Postpartum Depression
Brief Title: Effectiveness of Sertraline Alone and Interpersonal Psychotherapy Alone in Treating Women With Postpartum Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Caron Zlotnick, Director of Behavioral Medicine Research, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH074919 (NIH); R01MH074919 (NIH); R01MH074636 (NIH); DSIR 83-ATP
Record Dates: First submitted 2008-01-23; First posted 2008-01-28 (Estimated); Results first posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-07

CONDITIONS: Depression, Postpartum
Keywords: Postpartum; Depression; Medication Therapy; Zoloft; Sertraline; Interpersonal Psychotherapy
MeSH Terms: conditions — Depression, Postpartum; Depression | interventions — Sertraline; Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo) (Placebo Comparator): Participants receiving placebo pill with clinical management plus mothercrafting
  Interventions: Drug: Placebo; Behavioral: Clinical management; Behavioral: Mothercrafting
- 2 (Sertraline) (Active Comparator): Participants receiving active medication sertraline with clinical management plus mothercrafting
  Interventions: Drug: Sertraline; Behavioral: Clinical management; Behavioral: Mothercrafting
- 3 (IPT) (Active Comparator): Participants receiving interpersonal psychotherapy (IPT) alone
  Interventions: Behavioral: Interpersonal psychotherapy (IPT)

INTERVENTIONS:
Drug: Sertraline — Participants assigned to sertraline treatment will take 25 to 50 mg daily for Weeks 1 through 3, and dosage will be increased to 100 to 150 mg daily in Weeks 4 through 10. Participants will be titrated up to 200 mg daily at Week 11 for the final 2 weeks of treatment. In addition, at each week participants will receive specific "mother-crafting" techniques keyed to the baby's age and development. The mother-crafting component is aimed at providing relevant information to the mother about infant care.
  Other Names: Zoloft
  Arms: 2 (Sertraline)
Drug: Placebo — Participants taking the placebo will follow the same titration schedule as those taking sertraline. In addition, the participates will receive the same specific "mother-crafting" techniques as those taking sertraline.
  Arms: 1 (Placebo)
Behavioral: Interpersonal psychotherapy (IPT) — IPT will be administered in 13 individual 50-minute sessions over 13 weeks. These sessions will focus on improving relationships with others, setting goals, and increasing coping skills.
  Arms: 3 (IPT)
Behavioral: Clinical management — Clinical management includes treatment as usual for those receiving medication for depression.
  Arms: 1 (Placebo); 2 (Sertraline)
Behavioral: Mothercrafting — Mother-crafting techniques are keyed to the baby's age and development. The mother-crafting component is aimed at providing relevant information about infant care
  Arms: 1 (Placebo); 2 (Sertraline)

SUMMARY:
This study will evaluate the effectiveness of antidepressant medication alone and interpersonal psychotherapy alone in treating women with postpartum depression.

DETAILED DESCRIPTION:
Postpartum depression (PPD) occurs in approximately 13% of postpartum women. The impact of PPD is significant, including emotional distress for the woman as well as disturbances in infant development. Common signs of depression after childbirth may include anxiety, irritability, low energy, and lack of concern for self or infant. If left untreated, PPD may last for more than 1 year, causing strain on family life and the mother's relationship with her infant. Infants of depressed mothers are also at a higher risk for developmental delays, behavioral problems, and difficulty eating and sleeping. Despite the public health significance of PPD, relatively little research has been done to determine the most effective treatments. Specifically, there is a lack of research concerning the use of antidepressant medication for treating PPD. Interpersonal psychotherapy (IPT), which focuses on interpersonal issues related to depression, has been more thoroughly studied for the treatment for PPD, but it has not been compared to the other treatment. This study will evaluate the effectiveness of antidepressant medication alone and IPT alone in treating women with PPD.

Participation in this double-blind study will last 9 months. Participants will first undergo initial assessments, which include interviews about depressive symptoms, self-report forms about medical history, blood tests, and a pregnancy test. Participants will then be randomly assigned to one of three treatments: sertraline, placebo, or IPT. All three treatments will be administered over 13 weeks. Participants assigned to take sertraline or placebo will attend nine 30-minute sessions over the 13-week treatment period. During these sessions, participants will be administered the study medication and will be assisted with parenting issues and skills by a psychiatrist. Participants receiving IPT will attend weekly 50-minute sessions over the 13-week treatment period. These sessions will focus on improving relationships with others, setting goals, and increasing coping skills. All participants will also complete interviews and questionnaires about their depression once a month. Following the 13 weeks of treatment, participants will undergo follow-up assessments at Months 3 and 6 post-treatment. Follow-up assessments will repeat initial interviews and questionnaires and will include a form about the infant's nature.

ELIGIBILITY:
Inclusion Criteria:

* Primary DSM-IV diagnosis of major depressive disorder by clinical interview
* Score of greater than 12 on HAM-D
* Delivery of an infant within the 12 months prior to study entry
* Able to speak and read English sufficiently to complete the study procedures
* Willing to use effective birth control methods throughout the study

Exclusion Criteria:

* Woman whose infant has died prior to study entry
* Current or past diagnosis of bipolar disorder, schizophrenia or other psychotic disorder;
* Diagnosis of alcohol or drug abuse or dependence (except nicotine) or anorexia in the past year;
* Psychotic symptoms;
* Acute suicidal or homicidal risks;
* Women who have been on an antidepressant for more than 14 days prior to consent, (if less than 14 days and willing to taper off, will be eligible to continue once tapered off);
* Women on daily anxiolytic medication (i.e. benzodiazepine, buspirone) or daily psychoactive herbal preparation (St. John's Wort or Fish Oil) (if willing to discontinue these substances may be eligible once they have been tapered off);
* Medications taken PRN over the listed dose and frequency (women will still be eligible if they take: Lunesta/Eszopiclone 3 mg or less, up to 3 nights a week, Ambien/Zolpidem 5mg or less, Ambien CR 6.25 mg or less, up to 3 nights a week, Lorazepam or equivalent benzodiazepine dose: 0.5 mg up to 3 nights a week, Sonata/Zaleplon: 5 mg or less, up to 3 nights a week, Rozerem/Ramelteon: 8 mg or less, up to 3 nights a week);
* If they take antidepressants PRN for insomnia (eg: Desyrel/Trazodone, Elavil/Amitriptyline, Remeron/Mirtazapine;
* Ongoing concurrent psychotherapeutic treatment or psychotherapeutic treatment within the last month;
* Psychiatric symptoms requiring specialized psychiatric treatment;
* Significant medical disorder that would make sertraline treatment contra-indicated,
* Previous trial of IPT therapy with a certified IPT therapist or an adequate trial of sertraline (i.e. at least 8 weeks of at least 100 mg daily of sertraline).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2008-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caron Zlotnick, Principal Investigator — Women and Infants Hospital; Scott Stuart, MD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Women and Infants Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] O'Hara MW, Pearlstein T, Stuart S, Long JD, Mills JA, Zlotnick C. A placebo controlled treatment trial of sertraline and interpersonal psychotherapy for postpartum depression. J Affect Disord. 2019 Feb 15;245:524-532. doi: 10.1016/j.jad.2018.10.361. Epub 2018 Oct 31. PMID 30447565

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 (Placebo) | 2 (Sertraline) | 3 (IPT)
Started | 53 | 56 | 53
Completed | 44 | 38 | 43
Not Completed | 9 | 18 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 (Placebo) | 2 (Sertraline) | 3 (IPT) | Total
Number analyzed (Participants) | 53 | 56 | 53 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 56 | 53 | 162
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.28 (5.11) | 28.16 (5.63) | 26.26 (6.15) | 27.25 (5.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 56 | 53 | 162
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 14 | 13 | 44
  Not Hispanic or Latino | 36 | 41 | 40 | 117
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 10 | 24
  White | 31 | 36 | 32 | 99
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 14 | 13 | 10 | 37
Region of Enrollment [Number; unit: participants]
  United States | 53 | 56 | 53 | 162

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HAM-D)
Description: Measure total ranges from 0 to 50, with lower scores indicating better outcomes.
Time Frame: Measured at baseline; post-treatment; and Months 3 and 6 of follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 (Placebo) | 2 (Sertraline) | 3 (IPT)
Number analyzed (Participants) | 44 | 38 | 43
units on a scale
  Baseline | 22.0 (4.7) | 21.8 (4.7) | 22.0 (4.5)
  Post-Treatment | 8.8 (6.0) | 8.1 (7.1) | 8.2 (6.8)
  3-Month Follow-up | 6.7 (6.7) | 5.8 (6.5) | 7.3 (7.4)
  6-Month Follow-up | 6.5 (6.8) | 4.9 (5.7) | 6.1 (6.5)

2. Secondary Outcome: Depression Illness Severity Based on Beck Depression Inventory (BDI)
Description: Measure total ranges from 0 to 56, with lower scores indicating better outcomes.
Time Frame: Measured at baseline; post-treatment; and Months 3 and 6 of follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 (Placebo) | 2 (Sertraline) | 3 (IPT)
Number analyzed (Participants) | 44 | 38 | 43
units on a scale
  Baseline | 26.2 (7.7) | 27.0 (8.0) | 25.9 (8.3)
  Post-Treatment | 10.8 (11.5) | 10.0 (10.2) | 10.5 (10.2)
  3-Month Follow-up | 8.5 (8.7) | 7.3 (9.1) | 10.7 (11.0)
  6-Month Follow-up | 9.2 (10.0) | 5.1 (7.0) | 7.8 (8.8)

3. Secondary Outcome: Global Illness Severity Based on Clinical Global Impression (CGI) Scale
Description: Measure total ranges from 1 to 7, with lower scores indicating better outcomes.
Time Frame: Measured at baseline; post-treatment; and Months 3 and 6 of follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 (Placebo) | 2 (Sertraline) | 3 (IPT)
Number analyzed (Participants) | 44 | 38 | 43
units on a scale
  Baseline | 4.1 (0.7) | 4.0 (0.6) | 3.9 (0.8)
  Post-treatment | 2.1 (1.1) | 2.0 (1.2) | 2.0 (1.3)
  3-Month Follow-up | 1.9 (1.0) | 1.8 (1.2) | 2.0 (1.3)
  6-Month Follow-up | 1.7 (1.0) | 1.7 (1.1) | 1.8 (1.2)

4. Secondary Outcome: Social Functioning Based on Postpartum Adjustment Questionnaire (PPAQ)
Description: Measure total ranges from 1 to 5, with lower scores indicating better outcomes.
Time Frame: Measured at baseline; post-treatment; and Months 3 and 6 of follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 (Placebo) | 2 (Sertraline) | 3 (IPT)
Number analyzed (Participants) | 44 | 38 | 43
units on a scale
  Baseline | 2.7 (0.4) | 2.7 (0.4) | 2.6 (0.4)
  Post-Treatment | 2.4 (0.5) | 2.2 (0.4) | 2.3 (0.4)
  3-Month Follow-up | 2.3 (0.4) | 2.1 (0.4) | 2.3 (0.4)
  6-Month Follow-up | 2.3 (0.4) | 2.1 (0.4) | 2.2 (0.4)

5. Secondary Outcome: Hamilton Anxiety Rating Scale (HARS)
Description: Measure total ranges from 0 to 56, with lower scores indicating better outcomes.
Time Frame: Measured at baseline; post-treatment; and Months 3 and 6 of follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 (Placebo) | 2 (Sertraline) | 3 (IPT)
Number analyzed (Participants) | 44 | 38 | 43
units on a scale
  Baseline | 20.9 (6.6) | 20.3 (6.1) | 19.4 (6.2)
  Post-Treatment | 9.9 (8.0) | 9.4 (7.9) | 8.3 (9.0)
  3-Month Follow-up | 7.4 (7.8) | 6.6 (7.1) | 7.0 (7.5)
  6-Month Follow-up | 7.5 (8.4) | 6.2 (6.4) | 7.3 (8.3)

ADVERSE EVENTS:
Arm/Group | 1 (Placebo) | 2 (Sertraline) | 3 (IPT)
Serious Adverse Events (participants affected / at risk) | 7/53 | 8/56 | 8/53
Other Adverse Events (participants affected / at risk) | 20/53 | 19/56 | 16/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 (Placebo) (N=53) | 2 (Sertraline) (N=56) | 3 (IPT) (N=53)
Suicidal ideations or thoughts of self-harm (Psychiatric disorders) | 1 | 2 | 0
Attempted suicide (Psychiatric disorders) | 0 | 1 | 0
Infant hospitalized - bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Infant hospitalized - bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Participant hospitalized - gall bladder removal (Surgical and medical procedures) | 0 | 2 | 0
Participant hospitalized - kidney infection (Infections and infestations) | 0 | 0 | 1
Participant hospitalized - bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Worsening of neurovegetative symptoms (Psychiatric disorders) | 1 | 0 | 0
Infant hospitalized - dehydration, fever, vomiting (viral infection) (Infections and infestations) | 0 | 1 | 0
Participant hospitalized - hernia surgery (Surgical and medical procedures) | 0 | 0 | 1
Infant hospitalized - RSV (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Participant hospitalized - chest pain (General disorders) | 1 | 0 | 0
Participant hospitalized - kidney stone removal (Surgical and medical procedures) | 0 | 1 | 0
Infant hospitalized - croup cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Participant hospitalized - dehydration from excessive vomiting (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Participant hospitalized - hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Infant hospitalized - urinary infection and hand, foot, and mouth infection (Infections and infestations) | 1 | 0 | 0
Infant hospitalized - high fever (General disorders) | 1 | 0 | 0
Infant hospitalized - reaction to Enfamil (General disorders) | 0 | 0 | 1
Infant hospitalized - scheduled surgery for hydrocephalus (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 (Placebo) (N=53) | 2 (Sertraline) (N=56) | 3 (IPT) (N=53)
Participant reported experiencing headaches (General disorders) | 7 | 4 | 3
Participant reported experiencing insomnia (General disorders) | 2 | 5 | 3
Participant reported experiencing decreased libido (General disorders) | 7 | 2 | 0
Patient reported experiencing severe fatigue/sleepiness (General disorders) | 3 | 3 | 2
Worsening of symptoms (Psychiatric disorders) | 5 | 3 | 4 — Worsening of depressive or other psychiatric symptoms
Participant reported experiencing severe agitation (General disorders) | 2 | 1 | 3
Participant reported increased conflict with spouse or partner (Social circumstances) | 1 | 0 | 1
Patient reported experiencing delayed orgasm (Reproductive system and breast disorders) | 1 | 1 | 0
Patient reported hair loss (General disorders) | 0 | 1 | 0
Patient reported mild loss of appetite (General disorders) | 1 | 0 | 0
Participant ER visit - sprained ankle (Injury, poisoning and procedural complications) | 1 | 0 | 0
Participant reported ear infection (Infections and infestations) | 1 | 0 | 0
Participant reported experiencing toothaches (General disorders) | 1 | 0 | 0
Participant had 3 wisdom teeth removed (Surgical and medical procedures) | 1 | 0 | 0
Infant experiencing "mild" excessive drowsiness (General disorders) | 1 | 0 | 0
Participant reported that infant did not sleep (due to congestion) and is irritable (General disorders) | 1 | 0 | 0
Participant contracted ringworm from daughter (Infections and infestations) | 0 | 1 | 0
Participant screened positive on pregnancy test (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Participant reported experiencing dizziness/vertigo (General disorders) | 0 | 2 | 0
Participant reported fainting (General disorders) | 0 | 0 | 1
Infant had fever and diarrhea (General disorders) | 0 | 0 | 1
Participant had outpatient surgery on an existing hernia (Surgical and medical procedures) | 0 | 1 | 0
Participant injured eye while playing paintball - consulted doctor and healing well (Eye disorders) | 0 | 0 | 1
Participant ER visit - experiencing abdominal pain (General disorders) | 0 | 1 | 0
Participant reported experiencing itching and palpitations (General disorders) | 0 | 1 | 0 — resolved 1-2 days after stopping medication
Infant increased crying/fussiness, poor sleep, eating less, less frequent stool, less muscle tone (General disorders) | 0 | 1 | 0 — resolved when mother stopped breastfeeding for a day and discontinued use of study medication
Participant experienced rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Participant reported severe nervousness (General disorders) | 1 | 0 | 0
Participant experienced kidney infection (Infections and infestations) | 0 | 0 | 1
Increased conflict with other family and friends (Social circumstances) | 0 | 0 | 1
Infant experienced increased colic (General disorders) | 0 | 0 | 1
Separation from spouse (Social circumstances) | 0 | 0 | 1
Participant experienced sinus infection (Infections and infestations) | 1 | 0 | 0
Participant experienced pain due to having an IUD placed (General disorders) | 0 | 1 | 0
Participant ER visit - sinusitis (Infections and infestations) | 0 | 1 | 0
Participant diagnosed with 2 bulging discs causing back and leg pain (General disorders) | 0 | 0 | 1
Participant ER visit - shortness of breath, deemed likely to be anxiety related (Psychiatric disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No